CLINICAL TRIAL: NCT06029634
Title: Effects of T-bet B Cells in Persistent Virus Control After Discontinuance of NAs in CHB Patients
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, XueSong Liang, Dr, Changhai Hospital
Other Study IDs: T-bet B
Record Dates: First submitted 2023-08-28; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Chronic HBV Infection; Drug Withdrawal
Keywords: transcription factor bet; chronic hepatitis B; nucleotide analogs; function cure; B cell
MeSH Terms: conditions — Substance Withdrawal Syndrome; Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — pbmc
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- virologic breakthrough: CHB patients withdraw NAs with virologic breakthrough
  Interventions: Diagnostic Test: T-bet B cell
- virologic response: CHB patients withdraw NAs with virologic response
  Interventions: Diagnostic Test: T-bet B cell
- healthy group: The healthy (non-HBV infected) group completed a standard HBsAg vaccination scheduled before entering the study
  Interventions: Diagnostic Test: T-bet B cell

INTERVENTIONS:
Diagnostic Test: T-bet B cell — The frequency, function, and phenotype of T-bet B cells was tested

SUMMARY:
The immune mechanism of the nucleos(t)ide analogs (NAs) in inhibiting HBV replication effectively while having a low sustained virus control rate after drug withdrawal is unclear. B cell immunity and antibody response are the keys to prevent HBV reinfection and keep the virus under control. T-bet+ B, which can be regulated by IL-21, is a newly discovered major effector B cell in protection of pathogens and it is a main subtype of HBsAg-specific B cells. Thus, we suspect that T-bet+ B may play a role in ongoing controlling of the virus after withdraw of NAs in CHB patient. Based on our previous studies on CHB immunity, we use the RNAseq analyse, flow cytometry, and Elispot assay to analyze the frequency, function, and phenotype of B cells in CHB patients with different profiles after withdraw of NAs.

ELIGIBILITY:
Inclusion Criteria:

18 to 70 years old, no gender restriction, serum HBsAg positive than 6 months, can understand and sign informed consent, good compliance.

Exclusion Criteria:

coinfected with other hepatotropic virus such as hepatitis C virus,hepatitis D -virus,hepatitis E and hepatitis A etc; coinfected with HIV, markers such as ceruloplasmin, anti-nuclear antibodies and anti-mitochondrial antibodies for co-existent autoimmune and metabolic liver diseases were positive, with hepatocellular carcinoma(HCC) with uncontrollable extrehepatic disease, received glucocorticoid or other immune inhibitor therapy, pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CHB patients on NAs therapy
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
phenotype of B cells | PBMC were collected 0、4、12、24 week after withdraw the NAs
  CD19+cells were sorted from different samples, the frequency, function, and phenotype of B cells were analyzed.
B cell ELISPOT assay | Cells were stimulated with R-848 (1 μg/ml) and IL-2 (10 ng/ml) for 5 days at 37 °C to aid memory B cell differentiation
  Sorted B cell subsets were stimulated for 5 days following which B cell ELISPOT was conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Xuesong Liang, DR, Principal Investigator — Chaihai hospital
Locations (1):
- Changhai hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No